CLINICAL TRIAL: NCT06725940
Title: Clinical Study on the Evaluation of Neoadjuvant Therapy Efficacy in Breast Cancer Using PET/CT With Granzyme B Imaging Probe
Brief Title: GzmB-PET/CT to Evaluate Neoadjuvant Therapy Efficacy in Breast Cancer
Acronym: GzmB-PET4BC
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kunwei Shen, Professor, Shanghai Jiao Tong University School of Medicine
Other Study IDs: RJBC-GZMB
Record Dates: First submitted 2024-11-24; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Invasive
Keywords: breast cancer; Granzyme B; PET/CT; neoadjuvant treatment; pCR
MeSH Terms: conditions — Breast Neoplasms; Lipodystrophy, Congenital Generalized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Patient receiving 68Ga-GZMB PET/CT
  Interventions: Device: 68Ga-GZMB PET/CT

INTERVENTIONS:
Device: 68Ga-GZMB PET/CT — 68Ga-GZMB PET/CT

SUMMARY:
To explore the efficacy of 68Ga-GZMB PET/CT in assessing the response to neoadjuvant therapy for breast cancer, and to investigate the optimal SUVmax threshold of 68Ga-GZMB PET/CT for predicting pathological complete response (pCR), aiming to provide a new and effective means for accurately and non-invasively evaluating the efficacy of neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* age 16-65
* histologically confirmed unilateral primary invasive breast cancer
* Tumor size≥2cm, axillary lymph node positive, treated with neoadjuvant therapy
* complete clinical and histo-pathological information
* ECOG 0-1 within 10 days from the beginning of the study
* Normal Bone Marrow Reserve: White blood cell count ≥ 3.0×10^9/L, Neutrophil count ≥ 1.5×10^9/L, Hemoglobin level ≥ 90g/L; Platelet count (PLT) ≥ 80×10^9/L; Normal Liver and Kidney Function: Blood aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal, Total bilirubin ≤ 1.5 times the upper limit of normal, Serum creatinine ≤ 1.5 times the upper limit of normal, and Creatinine clearance rate > 50ml/min.
* The patient has good compliance with the planned treatment, understands the research procedures, and has signed a written informed consent form

Exclusion Criteria:

* bilateral or metastatic (stage IV) breast cancer
* There has been a history of other malignancies within the past 5 years, except for cured cervical carcinoma in situ and non-melanoma skin cancer
* Severe systemic infection or other uncontrolled diseases
* Patients with psychiatric disorders or those unable to comply with treatment due to other reasons
* Known allergy or intolerance to the drug or its excipients
* Having received cytotoxic chemotherapy, endocrine therapy, biological therapy, or radiotherapy for any reason in the past
* Patients who are pregnant or lactating, as well as patients of reproductive age who refuse to take appropriate contraceptive measures during the course of this trial.
* Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients receiving neoadjuvant treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Optimal SUVmax threshold of 68Ga-GZMB PET/CT for predicting pCR | through study completion, an average of 1 year
  Optimal SUVmax threshold of 68Ga-GZMB PET/CT for predicting pathological complete response after neoadjuvant therapy in breast cancer

SECONDARY OUTCOMES:
Sensitivity and specificity of 68Ga-GZMB PET/CT for pCR | through study completion, an average of 1 year
  Sensitivity and specificity of 68Ga-GZMB PET/CT in assessing pathological complete response after neoadjuvant therapy for breast cance
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 after 68Ga-GZMB PET/CT | through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 after 68Ga-GZMB PET/CT
Correlation between the efficacy of 68Ga-GZMB PET/CT in predicting pathological complete response and tumor-infiltrating lymphocytes | through study completion, an average of 1 year
  Correlation between the efficacy of 68Ga-GZMB PET/CT in predicting pathological complete response and tumor-infiltrating lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Xiaosong Chen, Principal Investigator — Shanghai Jiaotong University School of Medicine affiliated Ruijin Hospital
Locations (1):
- Shanghai Jiaotong University School of Medicine affiliated Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided